CLINICAL TRIAL: NCT02732964
Title: Perioperative Music for Patients Undergoing Scheduled Cesarean Delivery: Impact on Satisfaction, Anxiety, and Hemodynamic Response to Spinal Anesthesia
Brief Title: Impact of Music on Satisfaction, Anxiety, and Hemodynamics During Spinal Anesthesia for Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Michaela Kristina Farber, MD, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015P002043
Record Dates: First submitted 2016-04-01; First posted 2016-04-11 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Anxiety; Hypotension
Keywords: satisfaction
MeSH Terms: conditions — Anxiety Disorders; Hypotension; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): baseline hemodynamics and anxiety screen; no music
- Pandora Music (Experimental): A study investigator will create a station in the Pandora® music application based on the patient's preferred music genre or artist.
  Interventions: Other: Pandora Music
- Mozart Music (Experimental): A study investigator will turn on a playlist of pre-selected Mozart music.
  Interventions: Other: Mozart Music

INTERVENTIONS:
Other: Pandora Music — Patients enrolled will be exposed to Pandora music for 30 minutes prior to their spinal anesthesia and cesarean delivery, and throughout their surgery.
  Arms: Pandora Music
Other: Mozart Music — Patients enrolled will be exposed to Mozart music for 30 minutes prior to their spinal anesthesia and cesarean delivery, and throughout their surgery.
  Arms: Mozart Music

SUMMARY:
The aim of this study is to evaluate the effect of perioperative music on maternal anxiety, hemodynamic response to spinal anesthesia, postoperative pain medication requirement, and overall maternal satisfaction.

Investigators hypothesize that women exposed to perioperative music will have greater overall satisfaction with the delivery experience. Investigators also hypothesize that perioperative music will lower anxiety levels of women having a scheduled cesarean delivery, result in a less profound degree of spinal-induced hypotension prior to cesarean delivery, and result in a lower requirement of analgesics postpartum.

DETAILED DESCRIPTION:
Several studies have demonstrated that preoperative anxiety has been associated with more profound hypotension after spinal anesthesia for cesarean delivery. Music has been shown to have a positive impact on hemodynamic response and patient satisfaction.

To investigators knowledge, however, no studies have evaluated the effects of music during the perioperative period for cesarean delivery on patient satisfaction and hemodynamic responses.

The study will be conducted as a randomized unblended controlled trial with three study arms: control (no music), intervention - Pandora® (patient selected music), and intervention - Mozart (pre-selected relaxing music). Eligibility criteria include pregnant women, 18 years or older, scheduled for elective cesarean delivery under spinal anesthesia. Exclusion criteria include absolute contraindications of neuraxial anesthesia including patient refusal, uncorrected coagulopathy, infection at the skin site of epidural placement, increased intracranial pressure, or untreated hemodynamic instability. Patients in active labor, with impaired hearing, or who do not want to participate in the study will also be excluded. All subjects will be recruited from women admitted for scheduled cesarean delivery at Brigham and Women's Hospital. Investigators anticipate enrolling 150 patients, with 50 patients in each arm of the study.

Participation begins at the time of consultation on the day of surgery, and ends after the post-anesthesia check on postoperative day 1. After recruitment and consent, patients will be randomized using a computer-generated randomization scheme will be used to allocate patients to one of the arms of the study.

The three arms of the study are as follows:

1. Control group: baseline hemodynamics and anxiety screen; no music
2. Intervention group - Pandora: A study investigator will create a station in the Pandora® music application based on the patient's preferred music genre or artist.
3. Intervention group - Mozart: A study investigator will turn on a playlist of pre-selected Mozart music.

At the time of recruitment, patient demographic data and vitals signs will be collected. A baseline anxiety screen will be obtained (all groups) using the verbal analog scale (VAS) anxiety score and abbreviated State-Trait Anxiety Inventory (STAI) questionnaire. Thirty minutes prior to spinal anesthesia for cesarean delivery the designated music group will have music initiated, as described above. 30 minutes after completion of spinal placement, patient hemodynamics and vasopressor requirement (phenylephrine, ephedrine) will be evaluated by the co-investigator in 5 minute intervals. Thirty minutes after arrival in the post-anesthesia care unit postpartum, a postpartum anxiety screen will be obtained (all groups) using the VAS and STAI questionnaire. On postpartum day 1, all patients enrolled in this study will be evaluated within 24 hours of the spinal anesthetic.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* 8 years or older
* scheduled for elective cesarean delivery under spinal anesthesia.

Exclusion Criteria:

* absolute contraindications of neuraxial anesthesia including patient refusal
* uncorrected coagulopathy
* infection at the skin site of epidural placement
* increased intracranial pressure, or untreated hemodynamic instability.
* Patients in active labor, with impaired hearing, or who do not want to participate in the study will also be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-11; Primary Completion 2016-09 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
maternal anxiety level, VAS | prior to surgery
  assessed by VAS questionnaire
maternal anxiety level, VAS | 30 minutes after surgery
  assessed by VAS questionnaire

SECONDARY OUTCOMES:
Change in maternal blood pressure after spinal anesthesia induction , compared to baseline blood pressure | within 30 minutes of spinal placement
  nadir systolic arterial pressure within 30 minutes of spinal placement
maternal anxiety level, STAI | prior to surgery
  assessed by STAI questionnaire
maternal anxiety level, STAI | 30 minutes after surgery
  assessed by STAI questionnaire
Overall patient satisfaction, questionnaire | prior to surgery
  Assessed by questionnaire on postop day 1
Overall patient satisfaction, questionnaire | 30 minutes after surgery
  Assessed by questionnaire on postop day 1
Overall patient satisfaction, questionnaire | postoperative day 1
  Assessed by questionnaire on postop day 1
Overall patient satisfaction, pain control | prior to surgery
  Assessed by pain control/analgesic requirement on postop day 1
Overall patient satisfaction, pain control | 30 minutes after surgery
  Assessed by pain control/analgesic requirement on postop day 1
Overall patient satisfaction, pain control | postoperative day 1
  Assessed by pain control/analgesic requirement on postop day 1
Vasopressor requirement, phenylephrine | within 30 minutes of spinal placement
  utilization of phenylephrine, micrograms
Vasopressor requirement, ephedrine | within 30 minutes of spinal placement
  utilization of ephedrine, milligrams

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Drzymalski DM, Lumbreras-Marquez MI, Tsen LC, Camann WR, Farber MK. The effect of patient-selected or preselected music on anxiety during cesarean delivery: a randomized controlled trial. J Matern Fetal Neonatal Med. 2020 Dec;33(24):4062-4068. doi: 10.1080/14767058.2019.1594766. Epub 2019 Mar 27. PMID 30880522